CLINICAL TRIAL: NCT00594139
Title: An Open Label Multi-center Study of Augmentation Cystoplasty Using an Autologous Neo-Bladder Construct in Subjects With Non-Neurogenic Overactive Bladder and Urge Predominant Incontinence
Brief Title: Autologous Neo-Bladder Construct in Non-Neurogenic Overactive Bladder and Urge Predominant Incontinence
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Reprioritization of study programs
Sponsor: Tengion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNG-CL006
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Overactive Bladder
Keywords: non-neurogenic over active bladder; urge predominant incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Receipt of autologous neo-bladder construct
  Interventions: Biological: Autologous neobladder construct

INTERVENTIONS:
Biological: Autologous neobladder construct — provision of an autologous neo-bladder construct

SUMMARY:
Subjects with non-neurogenic over-active bladder will be enrolled. The hypothesis is that augmentation cystoplasty using an autologous neo-bladder construct will increase functional capacity and thereby reduce the number of micturition episodes per day in subjects with non-neurogenic over active bladder and urge predominant incontinence.

DETAILED DESCRIPTION:
Subjects with non-neurogenic over-active bladder and urge predominant incontinence who are intolerant to medical therapy or have persistence of symptoms despite medical therapy and require augmentation cystoplasty will be enrolled. The hypothesis is that augmentation cystoplasty using an autologous neo-bladder construct will increase functional capacity and thereby reduce the number of micturition episodes per day in subjects with non-neurogenic over active bladder and urge predominant incontinence.

ELIGIBILITY:
Inclusion Criteria:

* History of non-neurogenic overactive bladder for at least 12 months prior to study entry
* Intolerance to medical therapy or persistence of symptoms despite medical therapy

Exclusion Criteria:

* Subjects with stress incontinence or mixed incontinence where the predominant component is stress incontinence
* Use of Botulinum Toxin A injections into the bladder within the previous 6 months
* Presence of a neuromodulator
* Using catheterization as a way to control incontinence
* History of bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Mean number of micturitions per day | 12 months
Overall safety | 12 months

SECONDARY OUTCOMES:
Mean voided volumes, mean number of incontinent episodes, mean number of micturitions, cystometric capacity, detrusor pressure, end filling pressure and complaince | periodically within first 12 months as well as during long term follow up out to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tillinger, MD, Study Director — Tengion, Inc
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States